CLINICAL TRIAL: NCT06618430
Title: Evaluation Of DNA Methylation Pattern In Healthy, Sarcopenic, Obese And Sarcopenic Obese Older Women: A Cross-Sectional Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Other Study IDs: 73189623.6.0000.5659
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Sarcopenic Obesity; Sarcopenia; Obesity; Epigenesis, Genetic; Aging
Keywords: Sarcopenic Obesity; DNA Methylation; Aging
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood collection Blood samples will be collected in the morning after a 12-hour fast in EDTA tubes by experienced nurses. 5 ml of blood will be collected for analysis of biochemical markers (after centrifugation and separation of the plasma, it will be stored in a freezer at -80 °C for analysis) and genetic markers (DNA methylation, gene expression). Blood collection has minimal risk (Category 2; 45 CFR 46.110). All blood samples will be coded at the time of collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy older women: Older women who do not have sarcopenia, obesity or sarcopenic obesity.
  Interventions: Other: None (Observational Study)
- Older women with sarcopenia: Older women with sarcopenia, i.e. low handgrip strength and low muscle mass index.
  Interventions: Other: None (Observational Study)
- Older women with obesity: Older women with obesity
  Interventions: Other: None (Observational Study)
- Older women with sarcopenic obesity: Older women with sarcopenic obesity, i.e. low handgrip strength, low muscle mass index and high body mass index.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — None (Observational Study)

SUMMARY:
INTRODUCTION: Sarcopenic obesity (SO), a functional and clinical condition, is characterized by the coexistence of obesity, marked by excess fat mass and sarcopenia, characterized by reduced strength and muscle mass. SO is associated with a greater risk of health-related adverse clinical outcomes than older adults with obesity and sarcopenia alone. Aging is accompanied by numerous changes epigenetic. These aging-associated epigenetic changes include DNA methylation, histone modification, chromatin remodeling, non-coding RNA (ncRNA) regulation, and RNA modification. DNA methylation occurs at cytosines in CpG dinucleotides in the genome and undergoes changes with age in various human tissues. Furthermore, many genes can be hypermethylated or hypomethylated on CpG islands with the aging process. Soon, a broad exploration of candidate genes may provide insights into the pathogenesis of Sarcopenic obesity. Therefore, understanding how aging, specifically sarcopenia, obesity and Sarcopenic obesity, is regulated by epigenetic factors, favors the development of new treatment therapies. Thus, the objective will be to evaluate the epigenetic influence on sarcopenic obesity in older women. METHODS: This cross-sectional study will include 32 older women who will be classified as healthy, with sarcopenia, obesity and sarcopenic obesity living in the city of Ribeirão Preto - SP. The older adults will perform total and regional body scan using iDXA, anthropometric assessment, functional capacity tests, peripheral blood collection for analysis of biochemical markers and epigenetics. For statistical analysis will be used t test, ANOVA, linear regression models and Pearson correlation. Analyzes of the complete methylome will be performed using bioinformatics tools, including specific software. EXPECTED RESULTS: It is expected that there will be differences in the patterns of methylation and gene expression in the diseases analyzed. In addition, it is expected to clarify how epigenetic changes occur throughout this process.

DETAILED DESCRIPTION:
The sample size was calculated a priori, considering DNA methylation as the primary outcome, on an exploratory basis. The analyses were conducted using R software (https://www.r-project.org). For the calculation, an effect size of 0.65, alpha 0.05 and statistical power of 0.80 were used. Thus, a total of 32 participants will be included in the study (n = 8 in each group). The degree of methylation will be determined by measuring the amount of marker incorporated for each probe. The image intensities will be extracted using the Illumina Genome Studio 2011.1, Methylation module 1.9.0 software. The methylation score will be represented as a beta value (β) according to the fluorescence intensity ratio. Beta values can assume any value between 0 (unmethylated) and 1 (completely methylated). Subsequently, the image intensities will be extracted from the raw data (IDATS) using the Champ package for R (Statistical Computing, VIE, Austria). All genome-wide methylation data will be analyzed by t-test (within groups), followed by the Benjamini Hochberg test. Pathway enrichment analysis will be performed using WEBGestalt and Reactome. The normality of data distribution will be verified by the Shapiro Wilk test, and descriptive statistics will consist of mean and standard deviation values. ANOVA will be used to compare groups. Pearson correlations will be used to assess the correlation of DNA methylation patterns with phenotypic variables. Linear regression models will be applied to analyze the prediction of methylation pattern and selected variables. The multinomial logistic regression model will be used in the groups for association with telomere length adjusted for BMI, age, ALST). Statistical significance will be set at 5%, and all analyses will be performed using the Statistical Package for Social Sciences software (SPSS version 17.0 Inc. Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* body mass (menor 120 kg);
* sedentary (not practicing physical exercise for at least 3 months);
* not using vitamin or mineral supplements, anxiolytic medications, hypoglycemic agents with activity on cytochrome P450 (CYP450) enzymes;
* classified within the criteria for sarcopenic obesity, sarcopenia and obesity.

Exclusion Criteria:

* alcoholics;
* smokers;
* infectious diseases;
* coronary diseases;
* chronic kidney diseases and
* presenting a score ≤ 13 for the cognitive examination in the Mini-Mental State Examination (MMSE).

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants will be recruited through social media and on the website of the USP School of Physical Education and Sports (EEFERP/USP). Interested participants must register online and the researcher will then contact them by phone to schedule an interview.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Investigate whether the health condition (healthy, sarcopenic, obese or with sarcopenic obesity) promotes changes in DNA methylation | 1 day
  For this purpose, blood samples will be collected in the morning after 12 hours of fasting in EDTA tubes by experienced nurses. 5 ml of blood will be collected for analysis of biochemical markers and genetic markers (DNA methylation and gene expression). DNA extraction from peripheral blood will be performed with the AllPrepDNA/RNA/miRNA Universal kit (Qiagen), according to the instructions, using 200 µL of the extracted material. The quality of the extracted DNA will be assessed with the Greends DNA Quantification Reagent (Invitrogen, Carlsbad, CA, USA). After extraction, the samples will be stored in a freezer at -80°C for analysis. DNA will be bisulfite converted using the EZ DNA Methylation-Gold Conversion Kit (Zymo Research, CA, USA) according to the instructions, with conversion of unmethylated cytosine to uracil. Array-based specific DNA methylation analysis will be performed using the Infinium Human Methylation 850K (EPIC) Beadchip technology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, School of Physical Education and Sports of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No